CLINICAL TRIAL: NCT06649955
Title: Controlling Amyotrophic Lateral Sclerosis Motor Neuron Excitability Study
Acronym: CALM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PathMaker Neurosystems Inc. (Industry)
Collaborators: Beth Israel Deaconess Medical Center (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALS2; CDMRP-AL230079 (Other Grant/Funding Number: US Department of Defense)
Record Dates: First submitted 2024-10-14; First posted 2024-10-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: ALS - Amyotrophic Lateral Sclerosis
Keywords: ALS; Lou Gehrig's disease; Non-invasive; Multi-site direct current stimulation (multi-site DCS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Active MyoRegulator Treatment Arm (Experimental): 4 weeks of active MyoRegulator® device treatment three times per week then follow-up at 1 week, 1 month, 3 months, and optionally at 6 months following the end of treatment
  Interventions: Device: Multi-site direct current stimulation (DCS)

INTERVENTIONS:
Device: Multi-site direct current stimulation (DCS) — The MyoRegulator® treatment is a non-invasive intervention that suppresses motor neuron hyperexcitability and activates protein degradation pathways through the use of multi-site direct current stimulation (multi-site DCS).

SUMMARY:
Following completion of the ALS Early Feasibility Study of the MyoRegulator® device for treatment of ALS (NCT06165172), the CALM study will further assess the feasibility of the MyoRegulator® device to treat ALS in an expanded number of individuals with ALS. CALM will gather additional preliminary evidence of clinical safety and potential effectiveness in this patient population with a longer follow-up period and additional secondary endpoints in a single-arm study prior to commencing a larger sham-controlled pivotal trial.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS, Lou Gehrig's disease) is a progressive neurodegenerative disease that affects motor neurons in spinal cord and brain. ALS causes motor and cognitive function deficits and eventual death, typically within 2-5 years of diagnosis. There are at least 30,000 ALS patients in the United States and about 5,000 new diagnoses every year according to the Centers for Disease Control (CDC).

Central features of ALS pathology include the development of motor neuron hyperexcitability and the formation of protein aggregates in the cytoplasmic compartment of motor neurons and these are found across different ALS variants. The MyoRegulator® treatment is a non-invasive neuromodulation-based intervention that suppresses motor neuron hyperexcitability and activates protein degradation pathways through the use of multi-site direct current stimulation (multi-site DCS). Pre-clinical studies show that treatment using multi-site DCS effectively slows disease progression in transgenic mouse models of ALS. This is associated with improved motor function, preservation of motor neurons, and improved animal survival.

This clinical study is a non-significant risk (NSR), single-site, open-label investigation using the non-invasive multi-site DCS MyoRegulator® to evaluate the feasibility and safety of treatment with MyoRegulator® in individuals with ALS and to provide initial evidence of efficacy. The primary endpoint is feasibility and safety. Feasibility will be evaluated by recording and assessing the proportion potential participants who are enrolled from the total number of participants screened for the study, the ease of delivering treatment, the tolerability of study participants to the treatment, and the compliance of study participants with the study schedule and evaluations. Safety will be evaluated by recording the frequency and duration of any adverse events reported by study participants or observed by physical examination during or following treatment and throughout the study duration.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years of age inclusive
2. Sporadic or familial ALS diagnosed as clinically possible, probable, lab-supported probable, or definite ALS as defined by revised El Escorial criteria
3. Less than or equal to 3 years since ALS symptom onset
4. Slow Vital Capacity ≥ 50% of predicted capacity at the time of Screening as determined using a portable spirometer
5. For TTNCS: Median CMAP ≥ 1.5 mV
6. Willing to forgo botulinum toxin, phenol or alcohol injections, intrathecal baclofen, digitalis, and morphine for the study duration
7. Willing to refrain from participation in any other therapeutic clinical trial or investigational product for ALS for the duration of this study
8. Women must not be able to become pregnant (e.g., post-menopausal, surgically sterile, or using adequate birth control methods) for the duration of the study and 3 months after study completion.
9. Stable dose of rilutek (Riluzole), edaravone (Radicava), or tofersen (Qualsody) and oral medications for muscle spasms/cramps (e.g. mexiletine, quinine, quinidine, magnesium, gabapentin, oxcarbazepine, baclofen) for at least 30 days prior to the onset of participation in the study
10. ALS Functional Rating Score (ALSFRS-R) of greater than or equal to 35
11. Willing and able to give informed consent

Exclusion Criteria:

1. Study participants who are on permanent assisted ventilation (PAV) defined as >22h of noninvasive or invasive ventilation a day for > 7 consecutive days.
2. Study participants who have been diagnosed with ALS having only clinical bulbar involvement
3. Implanted intrathecal pump
4. Prior botulinum toxin injection(s) at any site within 12 weeks of study enrollment
5. Prior phenol or alcohol injections for spasticity within 6 months of study enrollment
6. Presence of potential tsDCS and/or TMS risk factors:

   1. Damaged skin at the stimulation sites (i.e., skin with ingrown hairs, acne, razor nicks, wounds that have not healed, recent scar tissue, broken skin, etc.)
   2. Presence of an electrically, magnetically or mechanically activated implant (including cardiac pacemaker) or any other electrically sensitive support system with the exception of loop recorders
   3. Ferromagnetic metal in the head, neck or any site of stimulation including, but not limited to, aneurysm clips, implanted medication pumps, implanted brain stimulators, pacemakers, cochlear implants, implanted metal prostheses or metal due to any injury; dental fillings are permitted. Jewelry must be removed during stimulation
   4. Seizures or unexplained spells of loss of consciousness during the previous 12 months
   5. Any cardiac abnormality that may be exacerbated by transthoracic electrical stimulation
   6. History of cord lesions or previous spinal surgery that may interfere with procedure as determined by the study MD
   7. History of intracranial brain lesions, cortical stroke or previous neurosurgery that may interfere with TMS (e.g., in regions to be stimulated for TMS evaluations) as reviewed and approved by the study MD
7. Any medical condition that would prevent the participant from being able to participate in the clinical outcome measures
8. Pregnant females, as determined by a pregnancy test at V1 (in females of child-bearing potential)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility of treating ALS patients using multi-site DCS | On treatment day and at each follow-up visit out to 3 months post-treatment
  The feasibility of treating ALS patients using multi-site DCS will be evaluated by determining the number of patients who can complete all of the study treatments at the target stimulation levels:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | On treatment day and at each follow-up visit out to 6 months post-treatment
  Safety will be evaluated by recording the frequency and duration of any adverse events reported by study participants or observed by physical examination during or following treatment and throughout the study duration, with particular attention to any device-related serious adverse events or unanticipated adverse events.

SECONDARY OUTCOMES:
ALS Functional Rating Scale (ALSFRS-R) | Just prior to treatment start at study week 1, after the last treatment at study week 4, then during follow-up at study weeks 8, 16, and 28
  The Revised (ALSFRS-R) is a clinician administered outcome measure that provides an evaluation of function in ALS patients. The ALSFRS-R measures 12 aspects of physical function, ranging from one's ability to swallow and use utensils to climbing stairs and breathing. Each function is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0.
Rasch Overall ALS Disability Scale (ROADS) | Just prior to treatment start at study week 1, after the last treatment at study week 4, then during follow-up at study weeks 8, 16, and 28
  ROADS is a patient-reported outcome measure used to evaluate functional abilities for activities of daily living in patients with ALS. ROADS is scored by assigning each of its 28 items a value of 0, 1, or 2:
  0: Unable to perform the task
  1. Able to perform the task with difficulty or with assistance
  2. Able to perform the task without difficulty ROADS then provides a normed total score that ranges from 0 to 146. The normed score is linearly weighted, meaning that a 1-point change represents a consistent and quantifiable measurement of disability. A 2-point change reflects twice the amount of disability.
ALS Assessment Questionnaire (ALSAQ-40) | Just prior to treatment at study week 1, then during follow-up at study weeks 4, 8, 16, and 28
  The ALSAQ-40 is a patient-reported, 40-item questionnaire that measures five areas of health status (domains) in patients with Amyotrophic Lateral Sclerosis (ALS) or other motor neuron diseases: 1) physical mobility; 2) activities of daily living and independence; 3) eating and drinking; 4) communication; 5), and emotional functioning.
  Each item on the ALSAQ-40 is scored using a 5-point Likert scale from 0 to 4. The sum of the item scores for each domain is divided by the maximum possible score for that domain, and then multiplied by 100. A lower score indicates a higher health-related quality of life (HRQoL).
Accurate Test of Limb Isometric Strength (ATLIS) | At baseline the day prior to treatment start, after the last treatment at study week 4, and at follow-up during weeks 8, 16, and 28
  The ATLIS machine will be used to measure any changes in isometric muscle strength in the study patients over the course of the study.
Threshold tracking nerve conduction studies (TTNCS) | At baseline the day prior to treatment start, after the last treatment at study week 4, and at follow-up during weeks 5, 8, 16, and 28
  TTNCS is used to assess spinal motor neuron excitability.
Measurement of cortical motor neuron excitabiity using Trans-cranial magnetic stimulation (TMS) | At baseline the day prior to treatment start, after the last treatment at study week 4, and at follow-up during weeks 5, 8 and 16.
  TMS is used to assess any changes in cortical motor neuron excitability throughout the study compared to baseline. This assessment involves evaluating the motor evoked potential (MEP) and the resting motor threshold (MT) using single-pulse TMS and evaluating intracortical excitability using a paired-pulse technique.
Slow Vital Capacity (SVC) | At baseline the day prior to treatment start, after the last treatment at study week 4 and at follow-up during weeks 5, 8, 16, and 28
  SVC is used to assess respiratory function.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No